CLINICAL TRIAL: NCT07068698
Title: The Effects of Thumb Manipulation on Hand Grip Strength, Hand Function, and Sensory Parameters
Brief Title: Effects of Thumb Manipulation on Hand Grip Strength, Function, and Sensation
Acronym: THUMBFUN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Asst. Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMT0010
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Thumb Manipulation; Hand Grip Strength; Hand Sensory Function; Hand Function in Healthy Individuals; Sensory Function
Keywords: Thumb manipulation; Chiropractic; Hand grip strength; Hand function; Healthy individuals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blinded to the group assignments to reduce measurement bias. Participants will be aware of their group allocation due to the nature of the intervention (the control group does not receive any treatment). The care providers performing the manipulation will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic Manipulation Group (CMG) (Experimental): Participants in this group will receive chiropractic manipulation specifically applied to the thumb. The intervention will be administered twice a week for 4 weeks by a trained physiotherapist experienced in manual therapy techniques. Each session will involve standardized manipulation techniques aimed at improving thumb mobility, hand grip strength, sensory function, and overall hand function. No additional interventions or therapies will be provided during the study period.
  Interventions: Other: Thumb Manipulation
- Control Group (CG) (No Intervention): Participants in the control group will not receive any intervention or treatment during the 4-week study period. They will continue their usual daily activities without any specific therapy applied. Outcome measurements will be conducted at the same time points as the intervention group to allow for comparison.

INTERVENTIONS:
Other: Thumb Manipulation — This intervention consists of chiropractic manipulation techniques applied specifically to the thumb joint. The manipulation will be performed by a trained physiotherapist twice weekly for 4 weeks. The procedure aims to improve thumb joint mobility, hand grip strength, sensory function, and overall hand function. Each session includes standardized manual therapy maneuvers targeting the thumb's range of motion and soft tissue mobility without the use of any devices or medications. The intervention differs from other manual therapies by focusing solely on the thumb region.
  Other Names: Chiropractic Thumb Manipulation; Manual Thumb Mobilization
  Arms: Chiropractic Manipulation Group (CMG)

SUMMARY:
This randomized controlled study will aim to investigate the effects of thumb manipulation on hand grip strength, function, and sensation in healthy individuals. A total of 60 volunteers aged between 18 and 50 years will be recruited from Ortadağ Special Education and Rehabilitation Center. Participants will be randomly assigned to either a chiropractic manipulation group (n=30) or a control group (n=30), with an equal distribution of males and females in each group. The intervention group will receive thumb manipulation twice weekly for 4 weeks, while the control group will not receive any intervention. Outcome measures will include two-point discrimination (assessed with a discriminator), hand grip strength (measured using a dynamometer), pinch strength (evaluated with a pinch meter), and hand function (measured by the Duruöz Hand Index). Statistical analyses will be performed with a significance level set at p<0.05. It is expected that participants in the manipulation group will show greater improvements in all measured parameters compared to the control group, suggesting a positive effect of thumb manipulation on hand-related sensorimotor functions in healthy individuals.

DETAILED DESCRIPTION:
This study will be designed as a randomized controlled clinical trial to evaluate the effects of thumb manipulation on hand grip strength, functional ability, and sensory parameters in healthy individuals. Sixty volunteers aged between 18 and 50 years will be recruited from Ortadağ Special Education and Rehabilitation Center. After anthropometric assessments, participants will be randomly assigned into two groups: a chiropractic manipulation group (n=30) and a control group (n=30), with equal numbers of males and females in each group.

The intervention group will undergo thumb manipulation performed by a trained physiotherapist twice a week for four weeks. The control group will not receive any intervention during this period. All participants will be evaluated at baseline, at the end of the 4-week intervention, and at follow-up.

Outcome measures will include:

Hand grip strength, measured using a hand dynamometer, Pinch strength, assessed with a pinch meter on the thumb, index, and middle fingers, Two-point discrimination, evaluated on the thumbs using a discriminator tool, Hand function, assessed using the Duruöz Hand Index. This study will aim to determine whether a short-term thumb manipulation protocol can lead to measurable improvements in sensory and motor functions of the hand in a healthy population. The findings may provide a basis for future research involving clinical populations with hand dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50
* Willing to participate in the study
* Have signed the informed consent form
* Able to use verbal and written communication skills

Exclusion Criteria:

* Having contraindications that may prevent manipulation
* Having a history of congenital or acquired orthopedic or neurological conditions affecting the upper extremity
* Having a history of rheumatological diseases
* Having a history of trauma or surgery affecting the upper extremity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-06 (Estimated); Primary Completion 2025-08-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
Duruoz Hand Index | T0 (Baseline, before intervention), T1 (Week 2 of intervention), and T2 (Week 4, end of intervention
  The Duruöz Hand Index is a validated self-reported questionnaire used to assess hand function and disability in daily activities. It includes 18 items covering various tasks such as dressing, hygiene, kitchen activities, and carrying objects. Each item is scored on a scale from 0 (no difficulty) to 5 (unable to perform), with higher scores indicating greater hand disability.
Two-Point Discrimination Test | T0 (Baseline, before intervention), T1 (Week 2 of intervention), and T2 (Week 4, end of intervention)
  The Two-Point Discrimination Test is used to evaluate sensory perception and tactile acuity. It measures the smallest distance at which two points of contact can be perceived as separate. In this study, the test will be applied to the thumb (right and left) using a standardized discriminator tool. Lower discrimination distances indicate better sensory perception. The test provides objective data on changes in cutaneous sensory function.
Pinchmeter | T0 (Baseline, before intervention), T1 (Week 2 of intervention), and T2 (Week 4, end of intervention)
  Pinch strength will be measured using a standardized pinchmeter to assess lateral, palmar, and tip-to-tip pinch strength in the thumb, index, and middle fingers of both hands. The test will provide quantitative data on fine motor strength and thumb function. Higher values indicate increased pinch strength. The measurement will be used to evaluate the effect of thumb manipulation on hand function.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA H HATIK, Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No